CLINICAL TRIAL: NCT01805960
Title: Canakinumab for the Prevention of Recurrences After Electrical Cardioversion in Patients With Persistent Atrial Fibrillation (CONVERT-AF) Trial - A Randomized Double Blind Placebo Controlled Study
Brief Title: Canakinumab for the Prevention of Recurrences After Electrical Cardioversion: CONVERT-AF
Acronym: CONVERT-AF
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CONVERT-AF Version5 22.01.2013
Record Dates: First submitted 2013-03-05; First posted 2013-03-06 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — canakinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Canakinumab (Experimental): 1 s.c. injection of canakinumab 150mg directly after cardioversion
  Interventions: Biological: Canakinumab
- Placebo (Placebo Comparator): 1 s.c. injection directly after cardioversion
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Canakinumab
  Arms: Canakinumab
Biological: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the efficacy of a single injection of Canakinumab on AF recurrences within 6 months after electrical cardioversion in patients with persistent AF.

ELIGIBILITY:
Inclusion Criteria:

* EKG-documented AF
* Undergoing electrical cardioversion
* C-reactive protein ≥1.25mg/L
* Age ≥ 50 years, women need to be postmenopausal

Exclusion Criteria:

* Undergoing urgent cardioversion because of medical instability
* AF persistence after cardioversion or AF recurrence before randomization
* Atrial flutter
* Severe renal failure (creatinine clearance <30 ml/min)
* Known active or recurrent hepatic disorder (including cirrhosis, hepatitis A, B or C, or Alanine transaminase/aspartate aminotransferase levels >3x ULN or total bilirubin >2x ULN)
* History of malignancy other than basal cell skin carcinoma
* Known intolerance or allergic reactions to canakinumab
* Use of amiodarone within the last 6 months
* Known HIV or any other immune compromised state including neutropenia or immunodeficiency
* History of ongoing, chronic or recurrent infectious disease
* History or evidence of active tuberculosis (TB) infection at Visit 1 or one of the risk factors for tuberculosis such as but not limited or exclusive to:

  * History of any of the following: residence in a congregate setting (e.g. jail or prison, homeless shelter, or chronic care facility), substance abuse (e.g. injection or noninjection), health-care workers with unprotected exposure to patients who are at high risk of TB or patients with TB disease before the identification and correct airborne precautions of the patient.
  * Close contact (i.e. share the same air space in a household or other enclosed environment for a prolonged period (days or weeks, not minutes or hours)) with a person with active pulmonary TB disease within the last 12 months.
  * Evidence of tuberculosis infection, at Visit 1, determined as defined by local guidelines/ local medical practice (see also below for determination of tuberculosis status). If presence of tuberculosis is established then treatment (according to local guidelines) must have been completed prior to randomization. Completion of treatment is determined by local TB guidelines or in the absence of such guidelines the following has to be demonstrated: TB has been treated adequately with antibiotics, cure can be demonstrated, and risk factors resulting in TB exposure and contracting TB have been removed (e.g. the patient does not live anymore in high TB exposure setting).
* Patients on systemic corticosteroids or other anti-inflammatory drugs other than non-steroidal anti-inflammatory drugs
* Patients on any biological drug targeting the immune system
* Acute coronary syndrome or acute stroke within 3 months
* History of heart failure hospitalization within 3 months
* Planned major surgery including planned coronary artery bypass grafting
* Women of childbearing potential
* Live vaccinations within 3 months prior to the randomization visit (visit 2) or live vaccinations planned during the trial.
* Life expectancy <1 year
* Inability to comply with the study protocol
* Previously enrolled in CONVERT-AF
* Patients who have received an investigational drug or device within 30 days of first visit.
* History of alcohol and/or substance abuse that could interfere with the conduct of the trial

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Recurrence of atrial fibrillation | 180 days

SECONDARY OUTCOMES:
Recurrence of atrial fibrillation | 90 days
Change in plasma levels of C-reactive protein | 180 days
Time to first redo cardioversion | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: David Conen, Prof., Principal Investigator — Cardiology, University Hospital Basel
Locations (5):
- University Heart Center Hamburg, Hamburg, Germany
- Switzerland (4):
  - Department of Medicine, University Hospital, Basel, Basel
  - HUG Geneve, Geneva
  - CHUV Lausanne, Lausanne
  - Kantonsspital St. Gallen, Sankt Gallen